CLINICAL TRIAL: NCT02536651
Title: Reliability and Validity of the Finnish Versions of the Visual Analogue Scale Foot and Ankle and the Lower Extremity Functional Scale
Brief Title: Reliability and Validity of the Finnish Visual Analogue Scale Foot and Ankle and the Lower Extremity Functional Scale
Status: Completed | Type: Observational
Sponsor: Helsinki University Central Hospital (Other)
Collaborators: Central Finland Hospital District (Other)
Responsible Party: Principal Investigator, Jussi Repo, Researcher, Helsinki University Central Hospital
Other Study IDs: 343/13/03/02/13/5
Record Dates: First submitted 2015-08-23; First posted 2015-09-01 (Estimated); Last update posted 2017-08-16 (Actual); Status verified 2017-08

CONDITIONS: Foot Diseases; Ankle Disease
Keywords: validation studies, patient-reported outcome measures
MeSH Terms: conditions — Foot Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Procedure: Ankle surgery — Plastic or orthopedic surgery of the ankle

SUMMARY:
There are no validated patient-reported outcome measures to assess lower extremity function in Finnish language. The present study aimed to 1)translate and culturally validate the Finnish versions of the Visual Analogue Scale Foot and Ankle and the Lower Extremity Functional Scale, and 2) study the psychometric properties of these two questionnaires

DETAILED DESCRIPTION:
This study assesses the reliability and validity of the Finnish versions of the Visual Analogue Scale Foot and Ankle and the Lower Extremity Functional Scale. The English versions were translated and trans-culturally adapted into Finnish language according to well accepted international translation guidelines. The psychometric properties are assessed by internal validity, intraclass correlation coefficient and test-retest reliability.

ELIGIBILITY:
Inclusion Criteria:

* Pathology of the foot and ankle and
* Surgery due to foot and ankle problems

Exclusion Criteria:

* Other than foot and ankle surgery
* age under 18 years

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who have undergone surgery due to foot and ankle pathology
Sampling Method: Non-Probability Sample
Enrollment: 120 (Actual)
Dates: Start 2014-09; Primary Completion 2015-08 (Actual); Study Completion 2015-08 (Actual)

PRIMARY OUTCOMES:
The validity of the Visual Analogue Scale Foot and Ankle and the Lower Extremity Functional Scale | 2 months to 10 years
  Assessment of the validity
The reliability of the Visual Analogue Scale Foot and Ankle and the Lower Extremity Functional Scale | 2 months to 10 years
  Assessment of the test-retest reliability

SECONDARY OUTCOMES:
Visual Analogue Scale Foot and Ankle questionnaire | 2 months to 10 years
  The questionnaire assesses function of the ankle
Lower Extremity Functional Scale questionnaire | 2 months to 10 years
  The questionnaire assesses function of the ankle
Kasari FIT (Function Intensity Time) index | 2 months to 10 years
  The questionnaire assesses the physical function level
The 15-Dimensions health-related quality of life instrument | 2 months to 10 years
  The questionnaire assesses
Visual Analogue Scales | 2 months to 10 years
  The Visual Analogue Scales assessed pain
Visual Analogue Scales | 2 months to 10 years
  The Visual Analogue Scales assessed functional capabilities

CONTACTS AND LOCATIONS:
Overall Officials: Erkki J Tukiainen, MD, PhD, Study Director — Helsinki University Hospital and University of Helsinki